CLINICAL TRIAL: NCT00050245
Title: Safety, Tolerability, and Efficacy of Rituximab in Patients With Anti-Glycoconjugate Antibody-Mediated Demyelinating Neuropathy: A Double-Blind Placebo-Controlled Randomized Trial
Brief Title: Rituximab to Treat Neuropathy With Anti-MAG Antibodies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030057; 03-N-0057
Record Dates: First submitted 2002-12-02; First posted 2002-12-03 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-17

CONDITIONS: Polyneuropathies
Keywords: Neuropathy; B Cells; Anti-MAG; Demyelination; MAG; RITUXAN; Monoclonal Antibodies; Retuximab; Demyelinating Neuropathy
MeSH Terms: conditions — Polyneuropathies; Demyelinating Diseases | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
This study will test the safety and effectiveness of the drug Rituximab in treating a nerve disease called MGUS (also known as neuropathy with anti-MAG antibodies). Patients with MGUS have an abnormal protein called monoclonal IgM immunoglobulin that attacks the myelin sheath (protective coating) of nerves, causing them to not function properly. The disease affects the nerves in the legs or arms, and patients have numbness, tingling, muscle weakness, and unsteady gait. There are no adequate treatments. Immunosuppressive drugs or human immunoglobulin infusions can produce mild and transient improvement, but the benefits of these therapies are not significant.

The abnormal immunoglobulin protein in MGUS is produced by white cells called B lymphocytes. Rituximab is approved to treat B cell lymphomas. Also, the drug showed promise in a recent study of patients with demyelinating neuropathy associated with production of antibodies from B lymphocytes directed against certain nerve proteins. Although the number of patients treated with Rituximab was small, the drug was well tolerated and caused significant improvement in several of the patients.

Patients 25 years of age and older with MGUS may be eligible for this 2-year study. Candidates will be screened with a medical history, physical and neurological examinations, and blood tests.

Participants will be randomly assigned to receive intravenous (through a vein) infusions of either Rituximab or placebo (a solution that looks like Rituximab but has no active ingredient) once a week for 4 consecutive weeks. In addition, they will undergo the following tests and procedures:

* Monthly follow-up visits following Rituximab treatment for repeat physical and neurological examinations, blood tests, muscle strength measurements, and review of signs and symptoms.
* Two sessions of lymphapheresis, one at the beginning of the study and one a year later-to collect lymphocytes. For this procedure, whole blood is drawn through a needle in an arm vein, much like donating a unit of blood. The blood then flows through a catheter (plastic tube) into a cell separating machine, where the white blood cells are extracted and removed. The red cells and plasma are then returned to the body through a needle in the other arm. The procedure takes about 60 to 90 minutes.
* Electrophysiologic studies (electromyography and nerve conduction testing) are done once at the beginning of the study and again one year later. For electromyography, a small needle is inserted into a few muscles and the patient is asked to relax or to contract the muscles. The electrical activity of the muscle cells is recorded and analyzed by a computer. For nerve conduction testing, nerves are stimulated through small wire electrodes attached to the skin and the response is recorded and analyzed.

If this study indicates that Rituximab is beneficial against MGUS, patients who were assigned to receive placebo during the trial will be offered treatment with Rituximab (four weekly infusions) at the end of the study.

DETAILED DESCRIPTION:
This study will examine the safety, tolerability, and efficacy of the humanized monoclonal antibody Rituximab to induce a clinical and serological remission in patients with IgM-anti-glycoconjugate antibody-mediated demyelinating neuropathy. Rituximab is a monoclonal antibody specific for the common B cell antigen CD20. Its administration depletes pre-B and mature B lymphocytes without altering neutrophils or hematopoietic stem cells. In humans with indolent B cell lymphomas, Rituximab can be safely administered, is well tolerated, promotes selective B cell depletion and lowers the serum IgM levels. Preliminary experience in some patients with demyelinating polyneuropathy and IgM-anti-glycolipid antibodies has shown that Rituximab was beneficial in improving the patient's symptoms and reducing the anti IgM antibody levels. In the present study we will examine in a placebo randomized trial the efficacy of Rituximab in patients with polyneuropathy related to IgM-anti-glycolipid antibodies. Twenty-six patients will be randomized to receive placebo or Rituximab given at four weekly intravenous infusions of 375 mg/M(2). The primary outcome will be based on changes in the monthly measurements of the neuropathy scores. The fine specificities of the IgM antibodies to various glycoconjugates or differences in the affinity binding to various antigens in neural membranes will be explored before and after treatment. It is anticipated that the study will: a) provide a new, immune-based and target-oriented therapy for patients with this neuropathy and b) examine the pathogenic role of these antibodies in the cause of the disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Research subjects will have documented disability of IgM anti-glycoconjugate antibody-mediated demyelinating neuropathy.

Neuropathy associated with IgM monoclonal immunoglobulins reactivate to MAG or other glycoconjugates.

Willingness and legal ability to give and sign informed study consent.

Willingness to travel to NIH for scheduled protocol studies and treatment.

Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.

Adequate bone marrow, renal, and liver function: ANC greater than 1000/mm3, BUN/Cr with normal range for age, AST or ALT less than 2 x of upper limit of normal.

EXCLUSION CRITERIA:

Immunosuppressive drug therapy at the time of or 6 months prior to enrollment. Specifically, candidates may not be taking prednisone, cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, anti-lymphocyte agents, cyclophosphamide, methotrexate, or other agents whose therapeutic effect is immunosuppressive or could provoke neuropathy as undesirable secondary effect.

Any medical or social condition that precludes follow-up visits.

Any active malignancy or any history of a hematogenous malignancy or lymphoma. Patients with melanoma will be excluded. Patients with primary, cutaneous basal cell or squamous cell cancers may be enrolled providing the lesions are treated prior to enrollment.

Coagulopathy or requirement for anticoagulation therapy that would contraindicate protocol.

Platelet count less than 100,000/mm(3).

Hemoglobin less than 7.0 mg/dl.

Any known immunodeficiency syndrome included HIV infection.

Any history of cardiac insufficiency, major vascular disease, or symptomatic coronary artery disease. Patients with cardiomyopathy grade III or IV by the New York Heart Classification will be excluded from this study.

Systemic edema or pulmonary edema.

Chronic hypotension (SBP less than 100 mm Hg).

Any condition that would likely increase the risk of protocol participation or confound the interpretation of the data including active infections.

Pregnancy. Serum pregnancy test will be performed and must be negative in all women of childbearing potential enrolled in the study.

History of active psychiatric disorder that may interfere with participation in the study.

Patients below the age of 25 because this neuropathy does not occur in such age groups.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-11-27; Study Completion 2007-10-17

PRIMARY OUTCOMES:
Changes in neurological performance using the INCAT scales.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dalakas MC, Quarles RH. Autoimmune ataxic neuropathies (sensory ganglionopathies): are glycolipids the responsible autoantigens? Ann Neurol. 1996 Apr;39(4):419-22. doi: 10.1002/ana.410390402. No abstract available. PMID 8619518